CLINICAL TRIAL: NCT04342871
Title: A Pilot Study Evaluating the Feasibility, Acceptability, and Preliminary Evidence of Efficacy of the Families Addressing Cancer Together (FACT) Intervention
Brief Title: An Evaluation of the Families Addressing Cancer Together (FACT) Intervention
Acronym: FACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2030
Record Dates: First submitted 2020-03-29; First posted 2020-04-13 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: Neoplasms; Cancer; Parenting; Communication; Parents; Parent-Child Relations
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Intervention Model Description: Because this is a pilot study, all participants will receive the same intervention and no blinding will take place
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FACT (Experimental): Patients will receive access to intervention materials.
  Interventions: Behavioral: FACT

INTERVENTIONS:
Behavioral: FACT — Customized communication guidance to help parents with cancer talk about their cancer with their children.

SUMMARY:
This is a pilot feasibility and acceptability study to inform the development and testing of a novel communication intervention to support parents in their communication with children about cancer. The research questions to be answered by this study are whether the intervention being tested can be feasible and acceptable, and provide preliminary estimates of improvement in parental psychological distress.

DETAILED DESCRIPTION:
This is a single-arm, single center pilot study using a pretest-posttest design to evaluate the feasibility and acceptability of a psychosocial intervention, Families Addressing Cancer Together (FACT). The purpose of the intervention is to decrease parental anxiety by facilitating parental communication about cancer with their children. The primary hypothesis being tested is that an intervention that assists parents with their communication needs with their children can be feasible, acceptable, and reduce parental psychological distress. Findings from this study will inform a future grant application to further test this intervention in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent reviewed and signed;
* Age equal to or above 18 years;
* Ability to understand and comply with study procedures;
* Be a parent, primary caregiver, or guardian of at least one child between the ages of 3-19 years old with whom the subject has regular contact. The child must have cognitive ability to understand verbal communication;
* Have a new or recurrent diagnosis of invasive solid tumor malignancy within the past 6 months or have a solid tumor cancer diagnosis with disease that is either stage IV or equivalent;
* Have a cancer diagnosis that is likely to require systemic anti-neoplastic therapy, non-office based surgical intervention, radiation therapy, or palliative care/hospice within the next three months.

Exclusion Criteria:

* Unable to complete self-report instruments due to illiteracy, neurologic illness, inability to speak or read English, or other causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Park, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - University of North Carolina Hospital, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park EM, Deal AM, Heiling HM, Jung A, Yopp JM, Bowers SM, Hanson LC, Song MK, Valle CG, Yi B, Cassidy A, Won H, Rosenstein DL. Families Addressing Cancer Together (FACT): feasibility and acceptability of a web-based psychosocial intervention for parents with cancer. Support Care Cancer. 2022 Oct;30(10):8301-8311. doi: 10.1007/s00520-022-07278-x. Epub 2022 Jul 13. PMID 35831719
- See also: UNC Lineberger Comprehensive Cancer Center — https://unclineberger.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from October 2020 to April 2021 in one center in North Carolina. Although 53 participants consented, 5 subjects did not complete the baseline assessment, and 2 subjects' clinical conditions did not allow them to complete the study requirements. Forty -six participants received the baseline intervention, 35 out of 46 participants completed the 2-week intervention, and 29 out of 35 participants completed the 12-week intervention.
Pre-assignment Details: All participants were assigned to receive the intervention after completing baseline assessments.
Period: Overall Study
Arm/Group | FACT
Started | 53
Completed | 29
Not Completed | 24
Not completed — Death | 4
Not completed — Clinical deterioration/illness progression | 2
Not completed — Did not complete baseline assessments | 5
Not completed — Lost to Follow-up | 13

BASELINE CHARACTERISTICS:
Population: Includes participants who provided informed consent and completed baseline assessments
Arm/Group | FACT
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.87 (7.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 39
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the Intervention Measured by the Study Visit Satisfaction Form FACT Was Helpful
Description: Acceptability of the intervention will be assessed through participants' satisfaction ratings used a study-specific satisfaction scale, "Families Addressing Cancer Together (FACT) satisfaction scale." Four-items (0=not at all, 3=very), higher scores indicate more satisfaction.
Time Frame: 14 days
Population: Participants who completed 2-week satisfaction assessment, reporting acceptability (Somewhat or very helpful) on 4-point scale
Measure: Count of Participants; unit: Participants
Groups:
- FACT Was Helpful: Patients will receive access to intervention materials.
  FACT: Customized communication guidance to help parents with cancer talk about their cancer with their children.
Arm/Group | FACT Was Helpful
Number analyzed (Participants) | 29
Participants
  Yes | 26
  No | 3

2. Primary Outcome: Acceptability of the Intervention Assessed Via Semi-structured Interviews
Description: Participants were interviewed about their experiences with the study intervention using semi-structured interviews. Parents' comments on the intervention "helped them feel more comfortable and prepared to talk with their children about their illness" were graded as participants overall intervention satisfaction.
Time Frame: 14 days
Population: Individuals who received intervention materials and participated in semi-structured feedback interview
Measure: Count of Participants; unit: Participants
Arm/Group | FACT
Number analyzed (Participants) | 10
Participants
  Intervention was satisfactory | 10
  Intervention was not satisfactory | 0

3. Primary Outcome: Acceptability of the Intervention Measured by the Study Visit Satisfaction Form-FACT Was Useful
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- FACT Was Useful: Patients will receive access to intervention materials.
  FACT: Customized communication guidance to help parents with cancer talk about their cancer with their children.
Arm/Group | FACT Was Useful
Number analyzed (Participants) | 29
Participants
  Yes | 26
  No | 3

4. Primary Outcome: Acceptability of the Intervention Measured by the Study Visit Satisfaction Form Content Was Important
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FACT Was Helpful
Number analyzed (Participants) | 29
Participants
  Yes | 27
  No | 2

5. Primary Outcome: Acceptability of the Intervention Measured by the Study Visit Satisfaction Form- Overall Satisfaction
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FACT Was Helpful
Number analyzed (Participants) | 29
Participants
  Yes | 27
  No | 2

6. Secondary Outcome: Feasibility of Screening
Description: The number of subjects who were screened, recruited, and retained in the study were reported.
Time Frame: Baseline
Population: Number of individuals who were assessed for eligibility and found to eligible
Measure: Count of Participants; unit: Participants
Arm/Group | FACT
Number analyzed (Participants) | 69
Participants
  Screened | 69
  Recruited/consented | 53
  Completed baseline intervention | 46
  Completed 2-week intervention | 35
  Completed 12-week intervention | 29

7. Secondary Outcome: Feasibility of Recruitment
Description: Number of patients who enroll in the study
Time Frame: Baseline
Population: Number of individuals eligible for participation who enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | FACT
Number analyzed (Participants) | 53
Participants
  Number who consented for participation | 53
  Number who completed baseline assessments to receive intervention | 46

8. Secondary Outcome: Communication Self-efficacy Measured by the Adapted Communication Self-Efficacy Scale
Description: Assess the change in patient's communication self-efficacy. The adapted Communication Self-Efficacy scale is a 9-item Visual Analogue Scale assessing parent's confidence in their ability to tell their child about parental medical illness. The score range is 0 to 100 with higher scores indicating higher confidence.
Time Frame: Baseline, 14 days, 84 days
Population: Participants who completed the Communication self-efficacy scale at baseline, 14 days, and 84 days.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Number of participants completed Baseline
- 14 Days: Number of participants completed at 14 days.
- 84 Days: Number of participants completed at 84 days.
Arm/Group | Baseline | 14 Days | 84 Days
Number analyzed (Participants) | 46 | 34 | 27
score on a scale | 78.8 (20.6) | 82.8 (20.2) | 82.8 (23.5)
Statistical Analysis 1: Comparison: Baseline; Test type: Other — Pre-post comparison from baseline to 2-weeks post-intervention; p = 0.2, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Through study completion, an average of six months
Arm/Group | FACT
All-Cause Mortality (participants affected / at risk) | 4/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT04342871/Prot_SAP_000.pdf